CLINICAL TRIAL: NCT06311877
Title: Effects of Flavor Modification for Management of Radiation Induced Dysgeusia in Head and Neck Cancer Patients
Brief Title: Effects of Flavor Modification for Management of Radiation Induced Dysgeusia
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Responsible Party: Principal Investigator, Jennifer Larsson, Speech-Language Pathologist, University of South Florida
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6795
Record Dates: First submitted 2024-03-06; First posted 2024-03-15 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Dysgeusia
MeSH Terms: conditions — Dysgeusia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group given mBerry tablet (Experimental): For the experiment group, the clinician will be providing participant with daily 0.4 gram mBerry tablets (total of 112 tablets) to consume twice a day (for two meals) over an 8-week period. The participant will be provided with a log form to track mBerry use for the two meals each day for the 8-week period. They will be requested to bring log to each of the clinical visits which include bi-weekly taste assessments.
  Interventions: Dietary Supplement: mBerry
- Control group not receiving mBerry (Active Comparator): The control group will not be given a placebo. The control group will come to clinic for bi-weekly taste assessments.
  Interventions: Other: No intervention

INTERVENTIONS:
Dietary Supplement: mBerry — mBerry tablets (.4 grams), which contain protein within the miracle berry called miraculin.
  Arms: Experimental group given mBerry tablet
Other: No intervention — The control group will not received intervention.
  Arms: Control group not receiving mBerry

SUMMARY:
Intervention for dysgeusia in head and neck cancer patients undergoing radiation therapy. This research proposal aims to investigate potential benefits of mBerry in improving quality of life and nutritional outcome in head and neck cancer patients' post-radiation therapy. Our hypothesis is that cancer patients undergoing radiation therapy will benefit from use of miracle berry in treatment of dysgeusia.

DETAILED DESCRIPTION:
Dysgeusia, characterized by altered taste, is a common side effect of radiation used in oropharyngeal cancer treatment. Radiation affects taste buds, leading to issues like loss of appetite, malnutrition, dependence on feeding tubes, dysphagia, and impacts social and overall quality of life. Patients often report bitter, metallic or no taste with food after radiation. Miracle berries, known for interacting with sweet taste receptors, could potentially transform acidic tastes into sweet ones.

The aim is to explore mBerry's potential in alleviating dysgeusia, aiding patients in achieving better nutritional status and quality of life.This study includes the use of mBerry tablets, which contain protein within the miracle berry called miraculin, for the treatment of radiation-induced dysgeusia. mBerry is not approved by the Food and Drug Administration (FDA) for the treatment of radiation-induced dysgeusia. It is being used as part of this research study to find out if mBerry tablets improve taste outcomes among head and neck cancer patients after radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years
* Diagnosis of mandibular cancer, tonsillar cancer, and lingual cancer
* Receiving primary or adjuvant radiation therapy

Exclusion Criteria:

* Received a total glossectomy or total laryngectomy.
* Patients with allergies to peanut, latex, peach, or soy will be excluded as they are at increased risk of allergy to mBerry.
* Diagnosis of diabetes as well as prediabetic patients and those that are taking Metformin.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-09-08 (Actual); Primary Completion 2026-12-14 (Estimated); Study Completion 2027-04-14 (Estimated)

PRIMARY OUTCOMES:
5-Point Hedonic Rating Scale | Bi-weekly for 8 weeks
  Taste Test Scale used to assessing liking or preference of taste of a product. Dislike Very Much: Assigned a value of 1, this represents strong disliking. Dislike Slightly: Assigned a value of 2, indicating mild disliking. Neither Like nor Dislike: Assigned a value of 3, representing a neutral response.
  Like Slightly: Assigned a value of 4, indicating mild liking. Like Very Much: Assigned a value of 5, representing strong liking. The higher the number scored indicates the participants enjoyed the taste vs the lower the number participant liked the taste less.
Chemotherapy-induced Taste Alteration Scale (CITAS) | Bi-weekly for 8 weeks
  Perceived taste scale- Self- administered questionnaire of 18 items evaluated on a five-point. Using a Likert scale 1-5 (where 1 = no difficulty or absence of the disturbance and 5 = maximum difficulty or disturbance). Higher scores indicate more severe taste alterations.

SECONDARY OUTCOMES:
M.D. Anderson Dysphagia Inventory (MDADI) | Bi-weekly for 8 weeks
  Patient questionaire on swallow function. Scored on a scale score from 0 to 100. Lower the scores indicate a greater impact of dysphagia on the patients quality of life.
Functional Oral Intake Scale (FOIS) | Bi-weekly for 8 weeks
  Level of least restrictive diet- the higher the number the participant is able to eat by mouth the lesser of number the patient might be reliable on a feeding tube

OTHER OUTCOMES:
Patients weight measurement | Patients will be seen for 4 follow-up appointments in the 8 week time frame of the study. The patient will be weighed at the 1st and 4th follow-up visit.
  Weight

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Larsson, Principal Investigator — University of South Florida
Locations (1):
- University of South Florida, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No